CLINICAL TRIAL: NCT07260279
Title: Effect of Educational Sessions for Abortive Care on Maternity Nurses' Performance
Brief Title: Effect of an Educational Session for Abortive Women on Maternity Nurses' Practices
Acronym: EESAW-MNP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FNCU-NURSE-ABWOMEN-01
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Abortion; Practice; Maternity
Keywords: Abortion; Maternity nurses; Practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention Group (Experimental): All maternity nurses in this study received an educational intervention about abortion care practices, including pre-, immediate-, and post-abortion nursing care. The intervention aimed to improve nurses' practical skills through lectures, demonstrations, and discussions
  Interventions: Other: Educational Training Program on Abortion Care

INTERVENTIONS:
Other: Educational Training Program on Abortion Care — The educational intervention consisted of structured training sessions for maternity nurses focusing on abortion care practices, including lectures, demonstrations, and discussions to improve skills and practices

SUMMARY:
The goal of this study is to evaluate the effect of structured educational sessions for abortive women on the practices of maternity nurses.

The study aims to enhance nurses' clinical skills and patient care related to abortion management.

Participants will:

Attend educational sessions designed to improve nursing practices

Participate in activities and discussions led by experienced instructors

Be observed before and after the sessions to assess changes in clinical practices

The study will compare nursing practices before and after the intervention to determine the overall impact of the educational sessions on professional performance and patient care quality.

ELIGIBILITY:
Inclusion Criteria:

Registered maternity nurses working in obstetrics or gynecology departments.

Having at least one year of clinical experience in maternity or reproductive health units.

Willing to participate and provide informed consent.

Able to read and understand the educational materials provided.

Present at the workplace during the study and follow-up periods.

Not previously involved in similar abortion care training programs.

Exclusion Criteria:

Nurses on maternity or annual leave during the study period.

Administrative or non-clinical nursing staff.

Nurses with less than one year of professional experience.

Refusal to participate or withdrawal at any stage of the study.

Attendance of any concurrent external training on abortion or reproductive health during the study.

Incomplete participation in the educational intervention sessions.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in maternity nurses' practices regarding abortion care | Before and three months after the educational intervention
  The primary outcome will measure changes in maternity nurses' practices related to pre-, immediate-, and post-abortion care using an observational checklist and structured evaluation tool administered before and after the educational program.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided